CLINICAL TRIAL: NCT01258140
Title: Detection of Pulmonary Embolism With CT Pulmonary Angiography Using Reduced Contrast Medium and Radiation Dose: Comparison of 100 kVp and 80 kVp Protocols
Brief Title: Detection of Pulmonary Embolism With Low-dose CT Pulmonary Angiography
Acronym: REDOPED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Stanley Thomas Johnson Foundation, Bern, Switzerland (Unknown)
Responsible Party: Zsolt Szucs-Farkas, MD. PhD., Institute of Diagnostic, Interventional and Pediatric Radiology, University Hospital Bern
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 120/08
Record Dates: First submitted 2010-12-06; First posted 2010-12-10 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Embolism, Pulmonary
Keywords: CT angiography; radiation dose; contrast medium
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Patients examined with normal-dose Computed tomography pulmonary angiography
  Interventions: Radiation: Computed tomography pulmonary angiography
- 2 (Active Comparator): Patients examined with low-dose Computed tomography pulmonary angiography
  Interventions: Radiation: Computed tomography pulmonary angiography

INTERVENTIONS:
Radiation: Computed tomography pulmonary angiography — CT pulmonary angiography using iodinated contrast agent
  Arms: 1
Radiation: Computed tomography pulmonary angiography — CT pulmonary angiography using iodinated contrast agent
  Arms: 2

SUMMARY:
Computed tomography pulmonary angiography (CTPA) is the imaging method of choice to rule out acute pulmonary embolism based on its high sensitivity and specificity. Unfortunately, CTPA uses iodinated contrast media and can provoke contrast induced nephropathy. On the other hand, Computed tomography uses ionising radiation and is responsible for the half of the radiation exposure coming from medical sources.

Recent studies have proven that low-dose CTPA protocols using Computed tomography tube energy of 80 kVp and reduced volume of iodinated contrast media provide an increased vessel signal and good image quality at a significantly reduced patient exposure. However, there are no data on the sensitivity of low-kVp protocols.

The aim of this prospective randomized trial is to detect any difference between a normal-dose and a low-dose CTPA protocol in the diagnostic accuracy in the detection of acute pulmonary embolism (PE).

DETAILED DESCRIPTION:
Background

Pulmonary embolism (PE) is the third most common cause of death in the U.S., with at least 650,000 cases occurring annually. Its frequency is similar in Europe. With the new generation of multi-detector Computed tomography scanners it is possible to depict the pulmonary vascular tree with a single intravenous injection of iodinated contrast medium (CM) in one breath-hold. This non-invasive method can delineate pulmonary arteries to their third-fourth branches and its overall negative predictive value lies above 99%. Therefore, Computed tomography-angiography with multi-detector scanners (MDCTA) is nowadays the preferred modality over conventional angiography or nuclear scintigraphic ventilation-perfusion (V/Q) scanning of the lung to exclude acute Pulmonary embolism(PE).

Unfortunately, Computed tomography uses ionising radiation and is already the largest contributor of radiation dose to the population in the Western countries. Most recent reports suggest that 1.5 to 2% of all fatal cancers are induced by Computed tomography in the U.S, equalling 25,420 cases per year. Furthermore, the rate of young adults with suspected Pulmonary embolism (PE) repeatedly examined with Multidetector Computed Tomography Angiography (MDCTA) is growing. Therefore, policies to reduce patient exposure are becoming more important in order to reduce the risk of developing cancer in the patients´ later life. On the other hand, elderly patients, who often has an impaired renal function or diabetes, may develop contrast induced nephropathy after the application of iodinated contrast media in, which is one of the most common causes of renal failure. Reducing iodine load in this patient group can efficiently prevent nephropathy, saving patients from dialysis and reducing medical costs.

Computed tomography protocols using low x-ray tube potential are capable of lowering radiation exposure with simultaneous increase of signal from the contrasted vessels. Furthermore, the higher vessel signal makes a reduction of the injected iodinated contrast material possible. Thus, low-kVp pulmonary CTA is warranted for routine use not only in younger patients to reduce radiation dose but also in the elderly to reduce the risk of contrast induced nephropathy.

In 2007 we reduced the tube energy of our routine pulmonary Multidetector Computed Tomography Angiography (MDCTA) protocol from 120 to 100 kVp which significantly reduced radiation dose. Our experience in more than 200 patients and results from a simulation study show that 80 kVp CTPA protocols using reduced radiation exposure by 40% and reduced volume of the injected contrast material by 25% provide an excellent image quality and a very good delineation of PE in patients weighing up to 100 kg. However, there is no clinical evidence based from prospective trials on the impact of low-dose CTPA on the detection of PE. Therefore, a large scale prospective randomised study comparing 100 kVp and 80 kVp protocols in respect sensitivity and specificity is warranted.

Objective

Assessment of diagnostic accuracy with normal-dose and low-dose CTPA in the detection of pulmonary embolism and to show the non-inferiority of the latter.

Methods

This is a monocentric, prospective randomised clinical study involving 500 patients with suspected pulmonary embolism (PE) undergoing CT pulmonary angiography. Examinations are and will be only performed if they are clinically indicated.

All patients weighing less than 100 kg with indicated CT pulmonary angiography (CTPA)to exclude pulmonary embolism (PE) between September 2008 and December 2012 are regarded as possible study candidates. The patients, if eligible, are randomly examined using a normal-dose (100 kVp, 100 mAs, 100 mL CM @ 4 mL/s) or a low-dose (80 kVp, 150 mAs, 75 mL CM @ 3 mL/s) CTPA protocol. Patients characteristics are recorded. Studies will be analyzed for pulmonary embolism (PE) localization. Findings will be compared to results from sonography of the lower extremity veins and V/Q scan of the lungs, if these were indicated, to clinical scores (revised Geneva and Wells scores) and to PE related death/ medical evidence of pulmonary emboli(PE) in 90 days following CTPA.

ELIGIBILITY:
Inclusion Criteria:

* CTPA (CT pulmonary angiography) indicated based on clinical suspicion for pulmonary embolism
* patient's body weight < 100 kg
* informed consent form signed by patient

Exclusion Criteria:

* contraindication to iodinated contrast media
* pregnancy (if alternative imaging methods to exclude pulmonary embolism are available)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2008-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Evidence of Pulmonary Embolism (PE) on CT pulmonary angiography (CTPA) | 1 hour after CTPA
Accuracy of normal- and low-dose CTPA on composite reference standard | 90 days after CTPA

SECONDARY OUTCOMES:
Evidence of PE or deep venous thrombosis in 90 days following CTPA | 90 days after CTPA
PE-related death in 90 days after CTPA | 90 days after CTPA
Diagnostic confidence with normal- and low-dose CTPA | 2 months after recruitment of last patient
Radiation dose with both CTPA protocols | 2 months after recruitment of last patient

CONTACTS AND LOCATIONS:
Overall Officials: Zsolt Szucs-Farkas, MD, PhD, Principal Investigator — Institute of Diagnostic, Interventional and Pediatric Radiology, University Hospital Bern; Zsolt Szucs-Farkas, MD, PhD, Principal Investigator — Hospital Centre Biel, Vogelsang 84, CH-2502 Biel/Bienne
Locations (1):
- Institute of Diagnostic, Interventional and Pediatric Radiology, University Hospital Bern, Bern, Canton of Bern, Switzerland